CLINICAL TRIAL: NCT05229653
Title: Phase I Randomized, Single-blind, Placebo-controlled, Single-center Study of the Effect of Postoperative Administration of Single Dose Ketamine on Pain and Recovery After Robotic Removal of Endometriosis in Patients With Chronic Pelvic Pain
Brief Title: The Using Postoperative Ketamine and Exploring the Effect on Endometriosis Pain (UPKEEEP) Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to challenges reaching the target accrual for participation.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-01032
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis; Post Operative Pain
MeSH Terms: conditions — Endometriosis; Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low-Dose Ketamine (LDK) Treatment Group (Experimental)
  Interventions: Drug: Ketamine
- Control Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Participants in this arm will receive intravenously (IV) ketamine (0.6 mg/kg) while recovering in the post anesthesia care unit (PACU) on the day of the surgery after subject has been deemed to be stable (hemodynamically stable, awake). The study physician will administer the study intervention via an intravenous pump to deliver 0.6 mg/kg ketamine over at least 30 minutes.
  Arms: Low-Dose Ketamine (LDK) Treatment Group
Drug: Placebo — Participants in this arm will receive intravenously (IV) matching equal dose of placebo while recovering in the post anesthesia care unit (PACU) on the day of the surgery after subject has been deemed to be stable (hemodynamically stable, awake). The study physician will administer the study intervention via an intravenous pump to deliver equal volume saline over at least 30 minutes.
  Arms: Control Group

SUMMARY:
This is a randomized, single blinded, placebo-controlled trial to study the effectiveness of a subanesthetic dose (0.6 mg/kg) of ketamine versus placebo (saline) on postoperative pain and pain on adult female chronic pelvic pain patients undergoing robotic removal of endometriosis. The objective of the study is to explore the effect of a sub anesthetic dose of ketamine (0.6 mg/kg) vs. saline control on postoperative pain and recovery in chronic pelvic pain patients who have undergone robotic removal of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18 to 65 years old
2. Experiencing chronic pain, defined as experiencing moderate to severe pelvic pain for greater than 6 months
3. Scheduled to undergo robotic endometriosis removal surgery
4. Willing to comply with all study procedures and be available for the duration of the study.
5. Subject is medically stable.

Exclusion Criteria:

1. Cognitive impairment (by history) or clinical signs of altered mental status such as confusion, amnesia, disorientation, fluctuating levels of alertness, etc. that may interference with adherence to study procedures and/or participant safety.
2. Past ketamine or phencyclidine misuse or abuse
3. Schizophrenia or history of psychosis
4. Known sensitivity or allergy to ketamine
5. Liver or renal insufficiency.
6. History of uncontrolled hypertension, chest pain, cardiac arrythmia, stroke, head trauma, intracranial mass or hemorrhage or pressure, glaucoma, acute globe injury, uncontrolled thyroid disease, porphyria, or any other contraindication to ketamine. Use of lamotrigine, alfentanil, physostigmine, and 4-aminopyridine are contraindicated
7. Pregnancy or nursing women
8. Currently participating in another pain interventional trial
9. Unwillingness to give informed consent
10. Non-English-speaking patients as the EHP-30 instrument has only been licensed to NYULH in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Huang, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Kathy.haung@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (0) |  | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Pain Score on Visual Analogue Scale (VAS)
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Baseline
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Pelvic Pain Score on Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: Post-Operative Day (POD) 1
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pelvic Pain Score on Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: Post-Operative Day (POD) 27
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Pelvic Pain Score on Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: Post-Operative Day (POD) 55
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Pelvic Pain Score on Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: Post-Operative Day (POD) 83
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Score on General Anxiety Disorder-7 Screener (GAD-7)
Description: GAD-7 consists of 7 problems. Participants report how often they have been bothered by the 7 problems over the last 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day). The total score range is 0-21; the higher the score, the more severe the anxiety. 0-4=minimal anxiety, 5-9=mild, 10-14=moderate, 15-21=severe anxiety.
Time Frame: Baseline
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Score on General Anxiety Disorder-7 Screener (GAD-7)
Description: as for outcome 6
Time Frame: Post-Operative Day (POD) 1
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Score on General Anxiety Disorder-7 Screener (GAD-7)
Description: as for outcome 6
Time Frame: Post-Operative Day (POD) 27
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Score on General Anxiety Disorder-7 Screener (GAD-7)
Description: as for outcome 6
Time Frame: Post-Operative Day (POD) 55
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Score on General Anxiety Disorder-7 Screener (GAD-7)
Description: as for outcome 6
Time Frame: Post-Operative Day (POD) 83
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Score on Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: MADRS is a 10-item diagnostic questionnaire that psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a 0-6 scale, resulting in a total score range of 0-60. The higher the score, the more severe the depression.
Time Frame: Baseline
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Score on Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 11
Time Frame: Post-Operative Day (POD) 1
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Score on Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 11
Time Frame: Post-Operative Day (POD) 27
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Score on Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 11
Time Frame: Post-Operative Day (POD) 55
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Score on Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 11
Time Frame: Post-Operative Day (POD) 83
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Score on Endometriosis Health Profile-30 (EHP-30) Questionnaire
Description: A Health-Related Quality of Life (HRQoL) patient self-report tool used to measure the wide range of effects that endometriosis can have on patients' lives, including work, relationship with child/children, sexual relationship, feelings about medical profession, feelings about treatment, and feelings about infertility. The EHP-30 questions are asked regarding endometriosis in the previous 4 weeks and are answered on a 5-point Likert scale, where 0=never, 1=rarely, 2=sometimes, 3=often, and 4=always. Raw scores for the questions within a scale are summed and transformed to a 0-100 scale, with higher scores indicating worse HRQoL.
Time Frame: Baseline
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Score on Endometriosis Health Profile-30 (EHP-30) Questionnaire
Description: as for outcome 16
Time Frame: Post-Operative Day (POD) 1
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Score on Endometriosis Health Profile-30 (EHP-30) Questionnaire
Description: as for outcome 16
Time Frame: Post-Operative Day (POD) 27
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Score on Endometriosis Health Profile-30 (EHP-30) Questionnaire
Description: as for outcome 16
Time Frame: Post-Operative Day (POD) 55
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Score on Endometriosis Health Profile-30 (EHP-30) Questionnaire
Description: as for outcome 16
Time Frame: Post-Operative Day (POD) 83
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in Opioid Use
Description: Opioid use will be assessed through medical records and subject reports. Assessment of opiate use will be used to determine the opiate-sparing effects of the study drug.
Time Frame: Baseline, Post-Operative Day (POD) 83
Population: Only 1 participant was enrolled, participant was lost to follow up before any outcome measure data was collected.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: No participants were enrolled in the control arm.
Arm/Group | Low-Dose Ketamine (LDK) Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05229653/Prot_SAP_000.pdf